CLINICAL TRIAL: NCT05815888
Title: Evaluation of Perioperative Lung Ultrasound Scores (LUS) in Living Donor Nephrectomy Surgeries: A Prospective Observational Study
Brief Title: Evaluation of Perioperative Lung Ultrasound Scores (LUS) in Living Donor Nephrectomy Surgeries
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Emre Sertaç Bingül, Medical Doctor, Lecturer, Istanbul University
Other Study IDs: 2022/1879
Record Dates: First submitted 2023-01-30; First posted 2023-04-18 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Atelectasis, Postoperative; Pulmonary Complication
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Living donor nephrectomy patients: Patients who are scheduled for donor nephrectomy, and who will be operated in lateral position using laparoscopic techniques
  Interventions: Diagnostic Test: Lung Ultrasound Score

INTERVENTIONS:
Diagnostic Test: Lung Ultrasound Score — one hemithorax is consisted of 6 scanning zones. Each of them are evaluated via ultrasonography in terms of presence of vertical B lines (<4 B lines: 1 point; >3 B lines or thick B lines: 2 points; marked disturbance in pleural line: 3 points). Higher scores reflect worse outcomes such as atelectasis and consolidation, and totally 12 zones are evaluated.
  Three different time points are defined for LUS:
  T1: 5 minutes after orotracheal intubation T2: At the end of surgery, before extubation T3: 30 minutes after extubation, in postanesthesia care unit.
  DeltaT= T2LUS-T1LUS
  Blood gas analysis will be evaluated hourly throughout the surgery

SUMMARY:
Living donor nephrectomy surgeries can be performed in lateral position with laparoscopic technique which necessitates pneumoperitoneum. Considering the position and the pneumoperitoneum, lungs can be affected macroscopically. In this study, it is aimed to observe whether lungs are affected by the aforementioned entities. The hypothesis is based on possible deterioration of the lungs due to the physical features of laparoscopic nephrectomy. Lung Ultrasound Score (LUS) will be used to evaluate the actual condition of lungs. Accordingly, one hemithorax is consisted of 6 different zones, and depending on the existence of vertical B lines (that refers to atelectasis and consolidation) each zone is scored 0 to 3. Higher scores reflect worse lung conditions that is associated with the severity of atelectasis. The LUS will be performed at three time points that are 5 minutes after intubation (T1), at the end of surgery and before extubation (T2), and at 30th minute in the postanesthesia care unit (T3). Primary outcome will be the difference between T1 and T3, secondary outcomes will include perioperative blood gas analyses, intraoperative mechanic ventilator parameters, intraoperative total amount of fluid given, postoperative pulmonary complications.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* Kidney donors
* Nephrectomy for transplantation
* Laparoscopic surgery

Exclusion Criteria:

* Chronic obstructive pulmonary disease grade III-IV
* existing structural lung disease (eg. interstitial lung disease)
* Pulmonary hypertension (>25 mmHg)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult living donor nephrectomy patients who are scheduled for laparascopic nephrectomy
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-07-23 (Actual)

PRIMARY OUTCOMES:
The comparison of T1LUS (After intubation lung ultrasound score) T2LUS (Preextubation Lung ultrasound score) | Up to 6 hours
  In order to observe the change in lung ultrasound scores between presurgical and at the end of the surgery, T2LUS (Lung ultrasound score before extubation) and T1LUS (Lung ultrasound score 5 minutes after intubation) will be compared. (A value of 0 points LUS is the best condition of the lung with no consolidation or atelectasis. 36 points refer to worst condition of the lungs with atelectasis in all the zones.)

SECONDARY OUTCOMES:
Postoperative pulmonary complications | Up to Postoperative 7 days.
  Incidence of pulmonary complications such as respiratory failure, aspiration pneumonitis, pneumonia, acute respiratory distress syndrome, pneumothorax, atelectasis, bronchospasm.
Comparison of Postanesthesia care unit (PACU) Partial arterial oxygen pressure (PaO2) and Lung ultrasound score at 30 minutes after extubation | Up to 6 hours
  A blood gas analysis will be obtained in the 30th minute of postanesthesia care, and arterial partial oxygen pressure (mmHg) will be evaluated.
Comparison of Postanesthesia care unit (PACU) Partial arterial carbon dioxide pressure (PaCO2) and Lung ultrasound score at 30 minutes after extubation | Up to 6 hours
  A blood gas analysis will be obtained in the 30th minute of postanesthesia care, and arterial partial carbon dioxide pressure (mmHg) will be evaluated.
Comparison of total given fluid amount (milliliters) and preextubation lung ultrasound score (T2LUS) | Up to 6 hours
  In order to observe the relation between the crystalloid amount given (ml) and its relation to lungs' ultrasonographic condition, intraoperative total fluid amount given will be evaluated.
Comparison of Lung ultrasound scores (LUS) after intubation(T1) and 30th minute after (T3) extubation | Up to postoperative 1 hour
  To understand the effects of lateral position and pneumoperitoneum on the lungs in acute postoperative period, LUS measurement at T1 (5 minutes after intubation) and LUS measurement at T3 (30 minutes after extubation) will be compared. LUS score vary between 0 to 36 (0= worst, 36= best condition of the lungs).

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University Istanbul Faculty of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No